CLINICAL TRIAL: NCT05361538
Title: A Single-center, Prospective Randomized Controlled Study of Microwave Spherical Ablation and Traditional Microwave Ablation in the Treatment of Single Hepatocellular Carcinoma With a Diameter of ≤5cm
Brief Title: Study of Microwave Spherical Ablation and Traditional Microwave Ablation in Single Hepatocellular Carcinoma ≤5cm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Third Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: drjingxiang005
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Cancer; Microwave Ablation; Microwave Spherical Ablation; Prognosis
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA Group (Experimental): Use true circular microwave needle for ultrasound-guided thermal ablation in MSA （microwave spherical ablation） group.
  Interventions: Device: True circular microwave needle
- MWA Group (No Intervention): Use normal microwave needle for ultrasound-guided thermal ablation in MTA （microwave ablation） group.

INTERVENTIONS:
Device: True circular microwave needle — Use true circular microwave needle for thermal ablation
  Arms: MTA Group

SUMMARY:
Comparison of the progression-free survival, overall survival, local progression rates, complete ablation rates and the complications rate of MSA and traditional MWA in the treatment of single hepatocellular carcinoma with a diameter of ≤5cm.

DETAILED DESCRIPTION:
HCC is a serious threat to the health of people，Early treatment of HCC results in a good prognosis for patients. Microwave ablation (MWA) is an important method for the treatment of early HCC. The traditional MWA technology has a long diameter of the ablation foci which is much larger than the transverse diameter, so in order to obtain a sufficient transverse diameter, the long diameter is often too large beyond the tumor boundary. That will cause too much normal liver tissue is unnecessarily damaged, especially for patients with severe liver cirrhosis or patients with liver cirrhosis who have undergone liver resection. In addition, it is easy to cause damage to adjacent vital tissues and organs. Changes in tissue properties during ablation affect the stability of the microwave field, resulting in unpredictable ablation shapes, which may cause omissions during tumor ablation, especially in multiple overlapping ablation, resulting in incomplete ablation, or increasing the risk of local tumor progression after treatment. Microwave spherical ablation (MSA) technology is a new MWA technology. With the help of temperature control technology, field control technology and wave control technology, a single needle can produce predictable spherical ablation lesions. Theoretically, MSA can improve the controllability of the ablation foci, which is suitable for the purpose of conformal ablation of large tumors in clinical practice, thereby minimizing the damage of local thermal ablation to liver tissue and adjacent important organs. However, there are few reports on the comparison of the therapeutic effect of MSA and traditional MWA. This study intends to conduct a prospective randomized controlled study based on the two mature microwave treatment methods of MSA and traditional MWA ablation to explore the effectiveness and safety of MSA in clinical application, providing evidence-based medical evidence for the clinical application of MSA.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has high risk factors for HCC and was first diagnosed of HCC by by contrast-enhanced imaging (CECT/CEMRI/CEUS) and/or pathology ;
2. Age range 18 to 75 years old;
3. Single lesion with tumor diameter ≤5cm;
4. Patient refuses surgery and determines to undergo microwave ablation
5. Liver function Child Pugh A or B;
6. No extrahepatic metastasis or portal invasion;
7. Patient signs the informed consent.

Exclusion Criteria:

1. The lesion has received treatment, including local ablation therapy and TACE therapy, etc;
2. With portal vein invasion or extrahepatic metastases;
3. Patient is with severe cardiopulmonary insufficiency.
4. Patient is a pregnant or breastfeeding women.
5. Patient is considered to be unsuitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of progression-free survival between MSA and traditional MWA in HCC | 6 to 12 months
  Compare the time to tumor progression after therapy of MSA and traditional MWA in the treatment of single hepatocellular carcinoma with a diameter of ≤5 cm

SECONDARY OUTCOMES:
Comparison of the overall survival of MSA and traditional MWA in HCC | 12 to 60 months
  Compare the time to of all-cause mortality after therapy of MSA and traditional MWA in the treatment of single hepatocellular carcinoma with a diameter of ≤5cm
Comparison of local progression rates of MSA and traditional MWA in HCC | 6 to 12 months
  Local progression was defined as new lesions with hyperenhancement in the arterial phase and low enhancement in the portal or delayed phase found adjacent to the ablation lesion (≤5 mm) during follow-up. Compare the local progression rates after therapy of MTA and traditional MWA in the treatment of single hepatocellular carcinoma with a diameter of ≤ 5 cm
Comparison of complete ablation rates of MSA and traditional MWA in HCC | 1 month
  Complete ablation was defined as the tumor showing no enhancement in three stages on contrast-enhanced imaging. Compare the rate of complete ablation after therapy of MTA and traditional MWA in the treatment of single hepatocellular carcinoma with a diameter of ≤5 cm
Comparison of the complications rate of MSA and traditional MWA in HCC | immediately
  Compare the rate of the complications during and after the therapy of MSA and traditional MWA in the treatment of patients with single hepatocellular carcinoma with a diameter of ≤5cm

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Jing, Study Director — Tianjin Third Central Hospital
Locations (1):
- Tianjin Third Central Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No